CLINICAL TRIAL: NCT02422940
Title: An Extension Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of Dalfampridine Extended-Release Tablets. for the Treatment of Chronic Post-Ischemic Stroke Walking Deficits .
Brief Title: Study to Evaluate the Long-Term Safety, Tolerability and Efficacy of Dalfampridine.
Acronym: MILESTONE℠
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DALF-PS-1029
Record Dates: First submitted 2015-04-14; First posted 2015-04-22 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Post-ischemic Stroke
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dalfampridine-ER 7.5 mg (Active Comparator): Dalfampridine-ER 7.5 mg tablets taken orally twice daily, approximately 12 hours apart.
  Subjects who received active treatment in the antecedent core study will retain the dose assignment to which they were initially randomized (7.5 mg or 10 mg dalfampridine-ER tablets). Subjects who received placebo in the core study will be randomly assigned to receive 7.5 mg or 10 mg dalfampridine-ER tablets in this extension study.
  Interventions: Drug: dalfampridine-ER 7.5 mg
- dalfampridine-ER 10 mg (Active Comparator): Dalfampridine-ER 10 mg tablets taken orally twice daily, approximately 12 hours apart.
  Subjects who received active treatment in the antecedent core study will retain the dose assignment to which they were initially randomized (7.5 mg or 10 mg dalfampridine-ER tablets). Subjects who received placebo in the core study will be randomly assigned to receive 7.5 mg or 10 mg dalfampridine-ER tablets in this extension study.
  Interventions: Drug: dalfampridine-ER 10 mg

INTERVENTIONS:
Drug: dalfampridine-ER 7.5 mg
  Arms: dalfampridine-ER 7.5 mg
Drug: dalfampridine-ER 10 mg
  Other Names: Ampyra™
  Arms: dalfampridine-ER 10 mg

SUMMARY:
This is an extension study to evaluate the long-term safety, tolerability, and efficacy of two dose strengths of dalfampridine-ER.

DETAILED DESCRIPTION:
This is an extension study to evaluate the long-term safety, tolerability, and efficacy of two dose strengths of dalfampridine-ER twice daily tablets when administered for at least 12 months to subjects with chronic post-ischemic stroke walking deficits who have completed the controlled, double-blind Study DALF-PS-1016.

ELIGIBILITY:
Key Inclusion Criteria:

* Completion of the DALF-PS-1016 study
* Providing informed consent to continue into the DALF-PS-1029 long-term extension study
* Sufficient ambulatory ability to independently complete the Two Minute Walk Test (2MinWT) and 10 Meter Walk Test (10MWT) at the time of enrollment into the extension study

Key Exclusion Criteria:

* Seizures, new onset strokes (or other significant neurological event precluding long-term continuation) occurring during the antecedent DALF-PS-1016 study
* Calculated creatinine clearance of ≤ 50 mL/minute at the time of enrollment into the long-term extension study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Roberts, MD, Study Director — Acorda Therapeutics
Locations (66):
- United States (62):
  - Acorda Site #117, Gilbert, Arizona
  - Acorda Site #109, Berkeley, California
  - Acorda Site #170, Carlsbad, California
  - Acorda Site #138, Long Beach, California
  - Acorda Site #105, Newport Beach, California
  - Acorda Site #142, Pasadena, California
  - Acorda Site #153, Sacramento, California
  - Acorda Site #151, San Diego, California
  - Acorda Site #163, San Diego, California
  - Acorda Site #124, Colorado Springs, Colorado
  - Acorda Site #110, Danbury, Connecticut
  - Acorda Site #149, Fairfield, Connecticut
  - Acorda Site #130, Stamford, Connecticut
  - Acorda Site #115, Atlantis, Florida
  - Acorda Site #119, Deerfield Beach, Florida
  - Acorda Site #147, Gainesville, Florida
  - Acorda Site #128, Hialeah, Florida
  - Acorda Site #184, Jacksonville, Florida
  - Acorda Site #103, Miami, Florida
  - Acorda Site #133, Miami, Florida
  - Acorda Site #161, Naples, Florida
  - Acorda Site #106, Tampa, Florida
  - Acorda Site #181, Honolulu, Hawaii
  - Acorda Site #171, Chicago, Illinois
  - Acorda Site #148, Avon, Indiana
  - Acorda Site #188, Fort Wayne, Indiana
  - Acorda Site #156, Franklin, Indiana
  - Acorda Site #146, Lexington, Kentucky
  - Acorda Site #150, New Orleans, Louisiana
  - Acorda Site #175, Fulton, Maryland
  - Acorda Site #136, Boston, Massachusetts
  - Acorda Site #121, Boston, Massachusetts
  - Acorda Site #123, East Lansing, Michigan
  - Acorda Site #164, Farmington Hills, Michigan
  - Acorda Site #159, Grand Rapids, Michigan
  - Acorda Site #101, Kansas City, Missouri
  - Acorda Site #111, Great Falls, Montana
  - Acorda Site #140, Reno, Nevada
  - Acorda Site #131, New Brunswick, New Jersey
  - Acorda Site #177, Stratford, New Jersey
  - Acorda Site #172, New York, New York
  - Acorda Site #179, Patchogue, New York
  - Acorda Site #114, White Plains, New York
  - Acorda Site #166, Chapel Hill, North Carolina
  - Acorda Site #167, Durham, North Carolina
  - Acorda Site #162, Mooresville, North Carolina
  - Acorda Site #154, Raleigh, North Carolina
  - Acorda Site #132, Winston-Salem, North Carolina
  - Acorda Site #137, Columbus, Ohio
  - Acorda Site #116, Dayton, Ohio
  - Acorda Site #152, Corvallis, Oregon
  - Acorda Site #168, Portland, Oregon
  - Acorda Site #126, Portland, Oregon
  - Acorda Site #122, Philadelphia, Pennsylvania
  - Acorda Site #144, Providence, Rhode Island
  - Acorda Site #157, Memphis, Tennessee
  - Acorda Site #113, Dallas, Texas
  - Acorda Site #165, Dallas, Texas
  - Acorda Site #108, Houston, Texas
  - Acorda Site #182, Falls Church, Virginia
  - Acorda Site #176, Richmond, Virginia
  - Acorda Site #107, Spokane, Washington
- Canada (4):
  - Acorda Site #203, Fredericton, New Brunswick
  - Acorda Site #202, Halifax, Nova Scotia
  - Acorda Site #201, Greenfield Park, Quebec
  - Acorda Site #204, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg tablets taken orally twice daily, approximately 12 hours apart.
  Subjects who received active treatment in the antecedent core study will retain the dose assignment to which they were initially randomized (7.5 mg or 10 mg dalfampridine-ER tablets). Subjects who received placebo in the core study will be randomly assigned to receive 7.5 mg or 10 mg dalfampridine-ER tablets in this extension study.
  dalfampridine-ER 7.5 mg
- Dalfampridine-ER 10 mg: Dalfampridine-ER 10 mg tablets taken orally twice daily, approximately 12 hours apart.
  Subjects who received active treatment in the antecedent core study will retain the dose assignment to which they were initially randomized (7.5 mg or 10 mg dalfampridine-ER tablets). Subjects who received placebo in the core study will be randomly assigned to receive 7.5 mg or 10 mg dalfampridine-ER tablets in this extension study.
  dalfampridine-ER 10 mg
Period: Overall Study
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Started | 152 | 142
Completed | 31 | 21
Not Completed | 121 | 121

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg | Total
Number analyzed (Participants) | 152 | 142 | 294
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 142 | 294
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.87) | 64.6 (10.32) | 63.3 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 104
  Male | 98 | 92 | 190
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 9 | 17
  United States | 144 | 133 | 277

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective Was to Evaluate Serious and Non-serious Adverse Events for Study Participants as a Measure of Safety and Tolerability of Dalfampridine ER (Extended Release) for at Least 12-months.
Description: This extension study was designed to evaluate long-term safety, tolerability, and efficacy of dalfampridine-ER (extended release) in adult subjects with chronic post-ischemic stroke walking deficits. Subjects who had completed the placebo-controlled DALF-PS-1016 core study were eligible to enroll regardless of whether they had received active drug or placebo in the core study.
Time Frame: up to 12 months
Population: The Safety Population of 293 subjects included all subjects who received at least one dose of study treatment.
  *One subject was randomized but discontinued the study prior to receiving double-blind study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 151 | 142
Participants
  Subjects with at Least One TEAE | 102 | 99
  Subjects with at Least One Serious TEAE | 14 | 8
  Subjects by Maximum Severity (Mild) | 45 | 45
  Subjects by Maximum Severity (Moderate) | 43 | 43
  Subjects by Maximum Severity (Severe) | 14 | 11
  Subjects with at least One TEAEA leading to Discon | 12 | 7
  Subjects who Died Due to a TEAE | 1 | 0

2. Secondary Outcome: Change From Baseline on the Two-Minute Walk Test (2MinWT)
Description: 2 Minute Walk Test (2MinWT) and Change from Baseline by Visit
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
Feet
  Baseline | 309.59 (132.956) | 297.41 (143.722)
  Visit 2 (Day 15) Actual Value: number analyzed (Participants) | 146 | 135
  Visit 2 (Day 15) Actual Value | 319.24 (135.072) | 312.08 (146.818)
  Visit 2 (Day 15) Change from Baseline: number analyzed (Participants) | 145 | 134
  Visit 2 (Day 15) Change from Baseline | 9.72 (34.898) | 14.27 (34.824)
  Visit 3 (Month 1) Actual Value: number analyzed (Participants) | 141 | 128
  Visit 3 (Month 1) Actual Value | 322.95 (136.511) | 317.96 (146.419)
  Visit 3 (Month 1) Change from Baseline: number analyzed (Participants) | 141 | 128
  Visit 3 (Month 1) Change from Baseline | 10.81 (40.457) | 14.48 (39.961)
  Visit 4 (Month 2) Actual Value: number analyzed (Participants) | 131 | 125
  Visit 4 (Month 2) Actual Value | 328.01 (139.437) | 318.98 (147.429)
  Visit 4 (Month 2) Change from Baseline: number analyzed (Participants) | 131 | 125
  Visit 4 (Month 2) Change from Baseline | 16.67 (34.512) | 17.48 (37.385)
  Visit 5 (Month 3) Actual Value: number analyzed (Participants) | 108 | 108
  Visit 5 (Month 3) Actual Value | 323.29 (136.815) | 331.77 (140.872)
  Visit 5 (Month 3) Change from Baseline: number analyzed (Participants) | 108 | 108
  Visit 5 (Month 3) Change from Baseline | 15.44 (41.635) | 16.99 (41.207)
  Visit 6 (Month 6) Actual Value: number analyzed (Participants) | 80 | 72
  Visit 6 (Month 6) Actual Value | 335.28 (128.117) | 321.28 (133.484)
  Visit 6 (Month 6) Change from Baseline: number analyzed (Participants) | 80 | 72
  Visit 6 (Month 6) Change from Baseline | 16.38 (38.767) | 72 (10.00)
  Visit 7 (Month 9) Actual Value: number analyzed (Participants) | 45 | 41
  Visit 7 (Month 9) Actual Value | 312.98 (136.536) | 342.24 (129.673)
  Visit 7 (Month 9) Change from Baseline: number analyzed (Participants) | 45 | 41
  Visit 7 (Month 9) Change from Baseline | 21.88 (45.327) | 19.25 (33.597)
  Visit 8 (Month 12) Actual Value: number analyzed (Participants) | 34 | 23
  Visit 8 (Month 12) Actual Value | 330.07 (144.749) | 360.90 (107.895)
  Visit 8 (Month 12) Change from Baseline: number analyzed (Participants) | 34 | 23
  Visit 8 (Month 12) Change from Baseline | 23.65 (50.899) | 19.98 (34.067)
  Final Visit - Actual Value: number analyzed (Participants) | 32 | 23
  Final Visit - Actual Value | 320.34 (136.425) | 318.48 (126.718)
  Final Visit - Change from Baseline: number analyzed (Participants) | 32 | 23
  Final Visit - Change from Baseline | 20.23 (50.991) | 9.88 (51.867)

3. Secondary Outcome: Change From Baseline on the 10 Meter Walk Test (10MWT)
Description: 10 Meter Walk Test (10MWT) and Change from Baseline by Visit
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: Meter /second
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
Meter /second
  Baseline | 0.92 (0.454) | 0.89 (0.472)
  Visit 2 (Day 15) Actual Value: number analyzed (Participants) | 145 | 135
  Visit 2 (Day 15) Actual Value | 0.97 (0.498) | 0.94 (0.494)
  Visit 2 (Day 15) Change from Baseline: number analyzed (Participants) | 145 | 135
  Visit 2 (Day 15) Change from Baseline | 0.05 (0.118) | 0.05 (0.124)
  Visit 3 (Month 1) Actual Value: number analyzed (Participants) | 140 | 127
  Visit 3 (Month 1) Actual Value | 0.96 (0.470) | 0.98 (0.494)
  Visit 3 (Month 1) Change from Baseline: number analyzed (Participants) | 140 | 127
  Visit 3 (Month 1) Change from Baseline | 0.03 (0.124) | 0.06 (0.122)
  Visit 4 (Month 2) Actual Value: number analyzed (Participants) | 131 | 125
  Visit 4 (Month 2) Actual Value | 0.99 (0.502) | 0.98 (0.503)
  Visit 4 (Month 2) Change from Baseline: number analyzed (Participants) | 131 | 125
  Visit 4 (Month 2) Change from Baseline | 0.06 (0.136) | 0.08 (0.134)
  Visit 5 (Month 3) Actual Value: number analyzed (Participants) | 108 | 108
  Visit 5 (Month 3) Actual Value | 0.95 (0.489) | 1.00 (0.488)
  Visit 5 (Month 3) Change from Baseline: number analyzed (Participants) | 108 | 108
  Visit 5 (Month 3) Change from Baseline | 0.05 (0.146) | 0.08 (0.167)
  Visit 6 (Month 6) Actual Value: number analyzed (Participants) | 80 | 71
  Visit 6 (Month 6) Actual Value | 1.01 (0.497) | 0.99 (0.456)
  Visit 6 (Month 6) Change from Baseline: number analyzed (Participants) | 80 | 71
  Visit 6 (Month 6) Change from Baseline | 0.06 (0.145) | 0.07 (0.124)
  Visit 7 (Month 9) Actual Value: number analyzed (Participants) | 45 | 40
  Visit 7 (Month 9) Actual Value | 0.99 (0.582) | 1.06 (0.400)
  Visit 7 (Month 9) Change from Baseline: number analyzed (Participants) | 45 | 40
  Visit 7 (Month 9) Change from Baseline | 0.08 (0.205) | 0.08 (0.145)
  Visit 8 (Month 12) Actual Value: number analyzed (Participants) | 34 | 23
  Visit 8 (Month 12) Actual Value | 1.05 (0.563) | 1.08 (0.414)
  Visit 8 (Month 12) Change from Baseline: number analyzed (Participants) | 34 | 23
  Visit 8 (Month 12) Change from Baseline | 0.07 (0.198) | 0.06 (0.238)
  Final Visit - Actual Value: number analyzed (Participants) | 32 | 23
  Final Visit - Actual Value | 1.04 (0.534) | 0.91 (0.425)
  Final Visit - Change from Baseline: number analyzed (Participants) | 32 | 23
  Final Visit - Change from Baseline | 0.04 (0.199) | -0.03 (0.263)

4. Secondary Outcome: Change From Baseline on the Timed up and Go (TUG) Test
Description: The TUG measures mobility and balance and can predict the risk of falls. This test, which was initially called the Get-up and Go test, is considered a measure of dynamic balance. The subject is asked to stand up from a chair, walk 10 feet at a comfortable pace, turn around and be seated. The Timed Up and Go (TUG) is measured in seconds. There will be one practice test and then the timed test. Only the timed test will be analyzed at each visit time point. Reciprocal transformation may be performed if the time values are markedly skewed.
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
Seconds
  Baseline | 17.92 (19.899) | 20.16 (18.587)
  Visit 2 (Day 15) Actual Value | 18.59 (30.461) | 19.82 (20.019)
  Visit 2 (Day 15) Change from Baseline | 0.67 (12.640) | -0.40 (4.844)
  Visit 3 (Month 1) Actual Value | 17.28 (21.165) | 18.76 (19.267)
  Visit 3 (Month 1) Change from Baseline | -0.59 (3.215) | -0.61 (7.329)
  Visit 4 (Month 2) Actual Value | 17.57 (22.351) | 18.49 (16.563)
  Visit 4 (Month 2) Change from Baseline | -0.45 (3.644) | -1.32 (4.816)
  Visit 5 (Month 3) Actual Value | 18.10 (26.829) | 17.39 (16.509)
  Visit 5 (Month 3) Change from Baseline | 0.05 (7.321) | -1.60 (4.323)
  Visit 6 (Month 6) Actual Value | 17.75 (31.394) | 17.07 (15.532)
  Visit 6 (Month 6) Change from Baseline | 0.33 (9.273) | -1.36 (4.740)
  Visit 7 (Month 9) Actual Value | 22.93 (39.918) | 15.85 (14.085)
  Visit 7 (Month 9) Change from Baseline | 1.66 (11.085) | -1.08 (3.452)
  Visit 8 (Month 12) Actual Value | 16.80 (13.724) | 15.17 (15.635)
  Visit 8 (Month 12) Change from Baseline | 0.33 (4.536) | -0.50 (2.606)
  Final Visit - Actual Value | 17.38 (15.967) | 19.21 (20.596)
  Final Visit - Change from Baseline | 1.34 (6.416) | 1.25 (6.914)

5. Secondary Outcome: Change From Baseline on the Walking Impact Scale (Walk-12)
Description: The Walk-12 is a 12-question questionnaire that asks subjects to rate limitations of their mobility during the preceding two weeks on a 5-point scale (from 1= not at all to 5=extremely). For each visit, the Walk-12 score will be calculated by summing the 12 components and transforming into a scale with a range of 0 to 100. A higher score indicates a greater degree of limitation in walking. A negative change indicates an improvement in walking. 0 = no limitation in mobility to 100 extreme limitation in mobility. Walk-12 Score = 100 * [(Mean of the 12 items) - 1]/(5-1)
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
units on a scale
  Baseline | 47.37 (26.933) | 49.78 (26.583)
  Visit 2 (Day 15) Actual Value: number analyzed (Participants) | 143 | 134
  Visit 2 (Day 15) Actual Value | 47.00 (25.860) | 45.95 (25.275)
  Visit 2 (Day 15) Change from Baseline: number analyzed (Participants) | 141 | 132
  Visit 2 (Day 15) Change from Baseline | -0.57 (13.081) | -3.92 (14.235)
  Visit 6 (Month 6) Actual Value: number analyzed (Participants) | 81 | 73
  Visit 6 (Month 6) Actual Value | 42.72 (23.649) | 48.14 (25.484)
  Visit 6 (Month 6) Change from Baseline: number analyzed (Participants) | 81 | 73
  Visit 6 (Month 6) Change from Baseline | -1.95 (13.247) | -2.40 (14.457)
  Visit 8 (Month 12) Actual Value: number analyzed (Participants) | 34 | 25
  Visit 8 (Month 12) Actual Value | 45.47 (23.405) | 49.67 (24.501)
  Visit 8 (Month 12) Change from Baseline: number analyzed (Participants) | 34 | 25
  Visit 8 (Month 12) Change from Baseline | -6.13 (16.047) | -5.75 (12.986)
  Final Visit - Actual Value: number analyzed (Participants) | 32 | 23
  Final Visit - Actual Value | 44.21 (24.976) | 49.00 (25.078)
  Final Visit - Change from Baseline: number analyzed (Participants) | 32 | 23
  Final Visit - Change from Baseline | -9.18 (17.097) | -1.90 (12.530)

6. Secondary Outcome: Change From Baseline on the Stroke Impact Scale (SIS)
Description: The SIS consists of 59 items grouped in 8 domains: strength, hand function, activities of daily living (ADL) / instrumental activities of daily living (IADL), mobility, communication, emotion, memory and thinking, and participation/role function. The subject is asked to rate the level of difficulty in performing each item in the preceding week. Each item is scored on a 5-point scale ranging from 1 (inability to complete the item) to 5 (no difficulty experienced at all). For each domain, the SIS score will be calculated by summing all the items within the domain and transforming into a scale with a range of 0 to 100 as follows: SIS Score = 100 * [(Actual raw score - Lowest possible raw score)/ (Highest possible raw score-Lowest possible raw score)].
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
score on a scale
  SIS ADL/IADL - Baseline | 71.8 (18.38) | 75.1 (16.56)
  SIS ADL/IADL Visit 6 Actual | 72.8 (18.57) | 77.0 (16.14)
  SIS ADL/IADL Visit 6 Change from Baseline | 0.4 (9.13) | -0.2 (8.99)
  SIS ADL/IADL Visit 8 Actual | 72.3 (18.64) | 73.8 (15.14)
  SIS ADL/IADL Visit 8 Change from Baseline | 1.7 (10.49) | -0.3 (8.35)
  SIS Communication - Baseline | 88.6 (16.76) | 88.3 (17.81)
  SIS Communication Visit 6 Actual | 88.7 (16.43) | 88.6 (15.38)
  SIS Communication Visit 6 Change from Baseline | -0.1 (9.85) | 0.3 (11.87)
  SIS Communication Visit 8 Actual | 83.6 (22.74) | 89.7 (16.47)
  SIS Communication Visit 8 Change from Baseline | -1.2 (12.33) | -2.5 (8.97)
  SIS Emotion - Baseline | 67.3 (13.08) | 68.9 (13.16)
  SIS Emotion Visit 6 Actual | 66.5 (12.88) | 65.7 (12.08)
  SIS Emotion Visit 6 Change from Baseline | -1.01 (15.56) | -2.7 (14.26)
  SIS Emotion Visit 8 Actual | 64.5 (14.94) | 67.0 (14.37)
  SIS Emotion Visit 8 Change from Baseline | -2.6 (12.77) | 3.8 (13.48)
  SIS Hand Function - Baseline | 45.9 (34.01) | 48.4 (34.79)
  SIS Hand Function Visit 6 Actual | 47.3 (34.81) | 52.3 (32.30)
  SIS Hand Function Visit 6 Change from Baseline | 4.6 (17.57) | 1.3 (14.51)
  SIS Hand Function Visit 8 Actual | 46.2 (34.66) | 54.0 (31.95)
  SIS Hand Function Visit 8 Change from Baseline | 4.3 (20.12) | 3.3 (16.40)
  SIS Memory & Thinking - Baseline | 82.8 (19.45) | 82.8 (19.91)
  SIS Memory & Thinking Visit 6 Actual | 84.0 (19.32) | 84.9 (17.35)
  SIS Memory & Thinking Visit 6 Change from Baseline | 0.9 (9.10) | 0.9 (10.86)
  SIS Memory & Thinking Visit 8 Actual | 80.7 (20.51) | 87.1 (17.83)
  SIS Memory & Thinking Visit 8 Change from Baseline | 0.5 (10.95) | -1.0 (12.39)
  SIS Mobility - Baseline | 71.7 (18.98) | 72.8 (19.07)
  SIS Mobility Visit 6 Actual | 74.5 (18.52) | 74.2 (18.59)
  SIS Mobility Visit 6 Change from Baseline | 1.4 (9.76) | -0.9 (11.58)
  SIS Mobility Visit 8 Actual | 70.8 (16.66) | 68.6 (19.46)
  SIS Mobility Visit 8 Change from Baseline | 3.5 (13.56) | -2.2 (11.17)
  SIS Participation - Baseline | 64.8 (26.08) | 68.8 (22.85)
  SIS Participation Visit 6 Actual | 69.6 (24.73) | 70.7 (21.95)
  SIS Participation Visit 6 Change from Baseline | 3.4 (20.03) | 1.4 (15.97)
  SIS Participation Visit 8 Actual | 65.3 (23.95) | 65.8 (24.65)
  SIS Participation Visit 8 Change from Baseline | 4.3 (18.86) | -3.1 (19.26)
  SIS Physical Dimension Score (SIS 16) - Baseline | 63.6 (10.01) | 64.5 (9.94)
  SIS Physical Dimension Visit 6 Actual | 65.1 (10.14) | 65.1 (9.66)
  SIS Physical Dim. Visit 6 Change from Baseline | 0.7 (5.13) | -0.6 (5.31)
  SIS Physical Dimension Visit 8 Actual | 64.0 (9.52) | 62.8 (9.72)
  SIS Physical Dim. Visit 8 Change from Baseline | 1.5 (6.73) | -1.3 (4.92)
  SIS Strength - Baseline | 53.4 (23.02) | 53.3 (22.34)
  SIS Strength Visit 6 Actual | 51.5 (24.46) | 52.8 (21.25)
  SIS Strength Visit 6 Change from Baseline | -0.9 (15.85) | 0.0 (19.45)
  SIS Strength Visit 8 Actual | 48.5 (19.16) | 51.8 (21.54)
  SIS Strength Visit 8 Change from Baseline | -1.1 (17.91) | -1.3 (22.27)
  Stroke Recovery - Baseline | 60.3 (21.42) | 65.0 (17.03)
  Stroke Recovery - Visit 6 Actual | 64.0 (20.72) | 66.4 (17.19)
  Stroke Recovery Visit 6 Change from Baseline | 2.8 (15.08) | 1.5 (12.08)
  Stroke Recovery Visit 8 Actual | 62.4 (22.16) | 67.4 (18.03)
  Stroke Recovery Visit 8 Change from Baseline | 0.6 (13.16) | 1.8 (13.32)

7. Secondary Outcome: Subject Global Impression (SGI)
Description: The Subject Global Impression (SGI) is single item measure of treatment response that asks the subject to rate the effects of the investigational drug on his or her overall walking ability using a 7 point scale ranging from 1 = "Terrible" to 7 = "Delighted."
Time Frame: Visit 8 (Month 12)
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke. These were the only participants to finish the SGI study due to study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 33 | 24
Participants
  7 - Delighted | 6 | 2
  6 - Pleased | 7 | 8
  5 - Somewhat Satisfied | 6 | 8
  4 - Neutral/Mixed | 12 | 5
  3 - Somewhat Dissatisfied | 1 | 0
  2 - Unhappy | 1 | 0
  1 - Terrible | 0 | 1

8. Secondary Outcome: Change From Baseline on the 12-item Health Survey (SF-12)
Description: The SF-12 v2 (4-week recall) is a general health-related quality-of-life profile measure consisting of 12 items. The SF-12 Physical Component Summary (PCS) and the Mental Component Summary (MCS) scores will be derived and normed to a general United States population for score algorithm. The normalized PCS and MCS scores will be calculated at baseline, Month 12, and subsequent visits.
  SF-12 is a Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Day 1, up to 12 months
Population: The study was conducted in patients with chronic walking deficits from an ischemic stroke.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 146 | 136
score on a scale
  MCS - Baseline | 54.2 (11.26) | 54.4 (10.00)
  MCS - Visit 8 - (Month 12) Actual | 50.5 (11.83) | 54.5 (11.60)
  MCS - Visit 8 - (Month 12) Change from Baseline | -4.3 (10.48) | -2.4 (9.28)
  PCS - Baseline | 36.2 (9.11) | 37.0 (8.64)
  PCS - Visit 8 - (Month 12) Actual | 37.3 (8.12) | 34.4 (10.55)
  PCS - Visit 8 - (Month 12) Change from Baseline | 2.7 (7.42) | -2.3 (7.50)

ADVERSE EVENTS:
Time Frame: Date collected within 1 year.
Description: The Safety Population of 293 subjects included all subjects who received at least one dose of study treatment.
  *One subject was randomized but discontinued the study prior to receiving double-blind study treatment.
Arm/Group | Dalfampridine-ER 7.5 mg | Dalfampridine-ER 10 mg
All-Cause Mortality (participants affected / at risk) | 1/151 | 0/142
Serious Adverse Events (participants affected / at risk) | 14/151 | 8/142
Other Adverse Events (participants affected / at risk) | 102/151 | 99/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalfampridine-ER 7.5 mg (N=151) | Dalfampridine-ER 10 mg (N=142)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Antrial Fibrillation (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Cellutiis (Infections and infestations) | 1 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Complex Partial Seizures (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalfampridine-ER 7.5 mg (N=151) | Dalfampridine-ER 10 mg (N=142)
Ear And Labyrinth Disorders (Ear and labyrinth disorders) | 4 | 3
Vertigo (Ear and labyrinth disorders) | 2 | 1
Eye Disorders (Eye disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 3 | 9
Diarrhea (Gastrointestinal disorders) | 4 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Gastro esophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 5 | 8
Gait Disturbance (General disorders) | 3 | 2
Malaise (General disorders) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 11
Nasopharyngitis (Infections and infestations) | 6 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 13 | 19
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Ligament Sprain (Injury, poisoning and procedural complications) | 4 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 3
Blood Creatinine Phosphokinase Increased (Investigations) | 4 | 1
Blood Creatinine Increased (Investigations) | 2 | 1
Gout (Metabolism and nutrition disorders) | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Headache (Nervous system disorders) | 6 | 7
Dizziness (Nervous system disorders) | 5 | 7
Balance Disorder (Nervous system disorders) | 1 | 4
Hypoesthesia (Nervous system disorders) | 0 | 4
Syncope (Nervous system disorders) | 3 | 1
Amnesia (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 2 | 1
Paresthesia (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 4 | 7
Anxiety (Psychiatric disorders) | 1 | 3
Hematuria (Renal and urinary disorders) | 1 | 3
Renal Cyst (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 6 | 5
Hematoma (Vascular disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 3 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Diastolic Dysfunction (Cardiac disorders) | 0 | 1
Dilatation Ventricular (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.